CLINICAL TRIAL: NCT00760318
Title: Prospective Double Blind Evaluation of Levetiracetam (Keppra) for the Treatment of Cervical Dystonia
Brief Title: Keppra for Cervical Dystonia
Acronym: Keppra
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decided to stop enrollment to review data.
Sponsor: University of South Florida (Other)
Responsible Party: Robert A. Hauser, MD, MBA, University of South Florida
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UCB Pharma- Keppra
Record Dates: First submitted 2008-09-24; First posted 2008-09-26 (Estimated); Last update posted 2018-11-23 (Actual); Status verified 2008-09

CONDITIONS: Cervical Dystonia
Keywords: cervical dystonia, keppra, botox, spasmodic torticollis
MeSH Terms: conditions — Torticollis | interventions — Levetiracetam

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Keppra — There will be flexible dose titration increasing by 250 mg per week for 12 weeks to a maximum of 3000 mg divided BID.
  Other Names: levetiracetam

SUMMARY:
The purpose of this study is to evaluate if there is an improved response in CD symptoms when Keppra is used as adjunctive therapy to Botox.

DETAILED DESCRIPTION:
Up to 40 patients with cervical dystonia and receiving intermittent Botox injections will be enrolled in the study. Patients will be evaluated at baseline 12-16 weeks following their prior set of Botox injections. Patients will be evaluated using the TWSTRS Cervical Dystonia Scale. Any oral medications for the treatment of cervical dystonia will be stable for at least four weeks and will continue unchanged throughout the study. Following Baseline evaluation, subjects will undergo their standard set of Botox injections. This will consist of the same dose and approximate placement as their prior set of injections. Subjects will then be randomized to LEV or placebo. They will begin oral study medication beginning with an LEV dose of 250 mg each evening or placebo. There will be flexible dose titration increasing by 250 mg per week for 12 weeks to a maximum of 3000 mg divided BID. The subjects will be on a stable dose of medication for weeks 12 to 16 (or to week 20 in subjects with sufficient improvement that they do not require Botox injections). Subjects will be evaluated at weeks 4,8,12, 16, 20 and 24. The primary efficacy outcome measure will be the difference in change in TWSTRS score from baseline to week 16. Patients may undergo Botox injections prior to the week 16 visit if it is medically necessary or if the subject indicates that they are experiencing intolerable discomfort. In these cases, final evaluation will be performed prior to Botox injection and their scores will be carried forward to endpoint. Those subjects who have sufficient improvement such that they don't require Botox injections at or by week 16 will be monitored on study medication for an additional four weeks. Following Botox injection or 20 weeks, subjects will undergo a two-week off titration of study medication. Secondary outcome measures will include difference in change in TWSTRS score from baseline to weeks 4, 8, 12, 16, 20 and 24 in patient-reported pain scale, Clinical Global Impression scale, Clinical Patient Improvement scale, patient reported disability scale, and length of time between injections. Adverse events will be recorded and described. Serious Adverse events will be reported to the FDA in writing within 15 calendar days of knowledge of the event with a copy sent to UCB and the USF Internal Review Board.

A comparison across groups of the number of subjects who require injections prior to week 16 will be undertaken. In addition, a comparison across groups of the number of subjects not requiring injections at week 16 will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Patients will have received their last Botox injections 12-16 weeks ago
* Any oral medications for cervical dystonia will be stable for 4 weeks and will continue throughout the study

Exclusion Criteria:

* Less than 21 years old
* Received Botox more than 16 weeks ago
* Not on a stable dose of oral medications for cervical dystonia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2005-11; Primary Completion 2007-10 (Actual); Study Completion 2007-10

PRIMARY OUTCOMES:
Primary endpoint will be the difference in change in TWSTRS score from baseline to week 16. | Week 16

SECONDARY OUTCOMES:
Secondary outcome measures will include difference in change in TWSTRS score from baseline to weeks 4, 8, 12, 16, 20, and 24 in patient-reported duration of benefit for their Botox injection, and length of time between injections. | Weeks 4, 8, 12, 16, 20, 24